CLINICAL TRIAL: NCT01931826
Title: Treatment of Schistosomal Portal Hypertension: Assessment of Efficacy of Endoscopic Therapy Alone or in the Combined With Surgical Procedure
Brief Title: Treatment Schistosomal Portal Hypertension: Efficacy of Endoscopy or Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Ciências da Saúde de Alagoas (Other)
Responsible Party: Principal Investigator, Celina Maria Costa Lacet, Doctor, Universidade Estadual de Ciências da Saúde de Alagoas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNCISAL-2012-Treatment PHS
Record Dates: First submitted 2013-03-15; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Schistosomiasis Mansoni; Portal Hypertension; Upper Gastrointestinal Bleeding
Keywords: Schistosomiasis; Surgical treatment; Endoscopic treatment
MeSH Terms: conditions — Schistosomiasis mansoni; Hypertension, Portal; Gastrointestinal Hemorrhage; Schistosomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic treatment alone (Active Comparator): 3 to 5 sessions of sclerotherapy till eradication of esophageal varices.
  Interventions: Procedure: Endoscopic treatment
- Total EGDS + endoscopy (Active Comparator): Esophagogastric devascularization with splenectomy followed by endoscopic sclerotherapy of esophageal varices 2 months postoperatively.
  Interventions: Procedure: Endoscopic treatment; Procedure: Total EGDS+ endoscopy

INTERVENTIONS:
Procedure: Endoscopic treatment — The presence of gastroesophageal varices was confirmed by fiberoptic esophagogastroduodenoscopy (EGD). In view of the experience of our service and local circumstances at the time of the study, the endoscopic treatment of choice was sclerotherapy, performed with a Teflon-sheathed metal needle. The sclerosing agent was 2.5% monoethanolamine oleate. Esophageal varices visible on EGD in the pre- and post-treatment period were classified as small, medium or large on the basis of criteria proposed by Paquet. All complications attributable to sclerotherapy were recorded.
Procedure: Total EGDS+ endoscopy — Esophagogastric devascularization with splenectomy followed by endoscopic sclerotherapy of esophageal varices 2 months postoperatively.
  Arms: Total EGDS + endoscopy

SUMMARY:
Upper gastrointestinal bleeding (UGIB) is a major cause of morbidity and mortality in patients with portal hypertension secondary to schistosomiasis mansoni. Taking into account the endemic nature of schistosomiasis mansoni in our region and the high morbidity and mortality directly associated with rupture of esophageal varices and UGIB in affected patients, we conducted a prospective randomized trial in patients with schistosomiasis and a history of bleeding esophageal varices. Its purpose was to assess the efficacy of endoscopic treatment alone compared with the efficacy of sclerotherapy preceded by a surgical treatment: Esophagogastric devascularization with splenectomy (EGDS).

DETAILED DESCRIPTION:
This was a prospective, randomized, single-center study carried out at the Department of Clinical and Surgical Gastroenterology of Hospital Universitário Professor Alberto Antunes, Universidade Federal de Alagoas (HU/UFAL). It was approved by the local Research Ethics Committee (protocol #98/0039-3, code 4010000-6) and all patients provided written informed consent prior to study enrollment. Patients who met relative criteria for exclusion received the current standard of care and follow-up and were analyzed as a third group in the study.

Over a two-year period, 79 patients were recruited for elective treatment of SPH. The criteria for selection were: a) an established diagnosis of hepatosplenic schistosomiasis as the cause of portal hypertension; b) a history of UGIB secondary to rupture of esophageal varices, with at least 20 days having elapsed since the most recent episode of bleeding; and c) age between 15 and 65 years.

The exclusion criteria were: chronic alcoholism, defined as an alcohol intake of ≥60 g/EtOH/day in men and ≥40 g/EtOH/day in women; evidence of decompensated liver disease of mixed etiology or of any chronic disease that contraindicated surgery were considered absolute exclusion criteria; the relative criteria for exclusion were altered hemostasis (platelet count < 50×109/L or INR > 1.5); presence of fundal varices on endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age between 15 and 65 years;
* an established diagnosis of hepatosplenic schistosomiasis as the cause of portal hypertension;
* a history of UGIB secondary to rupture of esophageal varices, with at least 20 days having elapsed since the most recent episode of bleeding.

Exclusion Criteria:

* Chronic alcoholism, defined as an alcohol intake of ≥60 g/EtOH/day in men and ≥40 g/EtOH/day in women;
* evidence of decompensated liver disease of mixed etiology or of any chronic disease that contraindicated surgery were considered absolute exclusion criteria;
* the relative criteria for exclusion were altered hemostasis (platelet count < 50×109/L or INR > 1.5);
* presence of fundal varices on endoscopy.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-01; Primary Completion 2005-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Sucess of treatment evaluated clinically by the absence of UGIB in the two years o follow-up. | 24 months
  Its purpose was to assess the efficacy of endoscopic treatment alone compared with the efficacy of sclerotherapy preceded by EGDS.

SECONDARY OUTCOMES:
Endoscopic evaluation of presence and grade of esophageal varices were made in both groups during the follow-up. | 24 months

OTHER OUTCOMES:
No other outcomes were evaluated. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Celina Lacet, Doctor, Principal Investigator — Universidade Estadual de Ciências da Saúde de Alagoas
Locations (1):
- Universidade Federal de Alagoas, Maceió, Alagoas, Brazil